CLINICAL TRIAL: NCT07030413
Title: Weaning From High Flow Nasal Oxygen in Acute Respiratory Failure : a Target Trial Emulation From Nouvelle-Aquitaine Health Data Warehouses
Brief Title: Weaning From High Flow Nasal Oxygen in Acute Respiratory Failure : a Target Trial Emulation
Acronym: HFNO-Weaning
Status: Active, not recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Collaborators: University Hospital, Bordeaux (Other); University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: HFNO-Weaning
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Failure With Hypoxia; Respiratory Failure, ICU; High-Flow Nasal Oxygen Therapy
Keywords: high-flow nasal oxygen therapy; acute hypoxemic respiratory failure; weaning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFNO weaning trial group: Patients who underwent at least one weaning trial from HFNO
- No HFNO weaning trial group: Patients who did not underwent HFNO weaning trial

SUMMARY:
Acute respiratory failure is a frequent reason for admission to the intensive care unit (ICU). It is associated with high healthcare consumption and mortality.

High-flow nasal oxygen (HFNO) improves comfort, reduces the risk of intubation and may reduce the risk of mortality in the most severe patients with acute hypoxemic respiratory failure compared with other oxygenation strategies. Therefore, HFNO is recommended as a first-line non-invasive oxygenation strategy in acute hypoxemic respiratory failure.

The timing of weaning patients from HFNO is complex. On the one hand, failure to wean from HFNO is associated with prolonged duration of HFNO and prolonged ICU stay. On the other hand, continued HFNO in patients ready to be weaned may unnecessarily prolong ICU stay and contribute to overwhelming of ICU capacities.

The overarching goal of this study is to identify the characteristics of patients in whom weaning from HFNO is not beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18)
* Admitted to participating ICUs
* Treated with HFNO at the attending physician's discretion for acute respiratory failure (defined as respiratory rate ≥ 25 breaths/min)

Exclusion Criteria:

* Prophylactic HFNO to prevent reintubation after extubation
* Noninvasive ventilation before HFNO initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ICU patients admitted to the 3 participating centers and treated with HFNO at the attending physician's discretion for acute respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital-free days at day 90 | 90 days
  The number of days alive out of hospital between pseudorandomization and D90. For patients who died, the hospital-free days at day 90 will be equal to 0.

SECONDARY OUTCOMES:
Duration of intensive care unit (ICU) stay | 90 days
  The number of days spent in the ICU
ICU mortality | 90 days
  The number (and proportion) of patients who died in the ICU
Survival at day 90 | 90 days
  The number (and proportion) of patients alive at day 90 from pseudorandomization

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - University Hospital Bordeaux, Bordeaux
  - University Hospital Limoges, Limoges
  - University Hospital Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available after reasonable request and it has been discussed among the steering committee.

REFERENCES:
- [Background] Rodriguez M, Thille AW, Boissier F, Veinstein A, Chatellier D, Robert R, Le Pape S, Frat JP, Coudroy R. Predictors of successful separation from high-flow nasal oxygen therapy in patients with acute respiratory failure: a retrospective monocenter study. Ann Intensive Care. 2019 Sep 11;9(1):101. doi: 10.1186/s13613-019-0578-8. PMID 31511996
- [Background] Oczkowski S, Ergan B, Bos L, Chatwin M, Ferrer M, Gregoretti C, Heunks L, Frat JP, Longhini F, Nava S, Navalesi P, Ozsancak Ugurlu A, Pisani L, Renda T, Thille AW, Winck JC, Windisch W, Tonia T, Boyd J, Sotgiu G, Scala R. ERS clinical practice guidelines: high-flow nasal cannula in acute respiratory failure. Eur Respir J. 2022 Apr 14;59(4):2101574. doi: 10.1183/13993003.01574-2021. Print 2022 Apr. PMID 34649974